CLINICAL TRIAL: NCT06859398
Title: Data Collection Study in Keratoconus, Utilizing Topography and Wavefront Aberrometry
Brief Title: KeratoConus Data Acquisition With Topography and Aberrometry
Acronym: KC-DATA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azalea Vision (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Az01
Record Dates: First submitted 2025-03-04; First posted 2025-03-05 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Corneal Ectasia; Keratoconus
Keywords: Keratoconus; Corneal ectasia; Wavefront aberrometry; Corneal topography; Scleral topography; Ocular topography; Irregular corneal condition
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Intervention Model Description: This study is considered as a data collection study. The data which will be collected within this study, is not collected per standard of care. Depending on the participating country, the study is considered interventional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Keratoconus and corneal ectasia (Other): wavefront aberrometry and topography measurement through Pentacam AXL Wave device
  Interventions: Other: Ocular Topography and Wavefront Aberrometry

INTERVENTIONS:
Other: Ocular Topography and Wavefront Aberrometry — Eyescan with Pentacam AXL Wave

SUMMARY:
This observational study aims to collect real-world wavefront aberrometry and corneal/scleral topography data from individuals with keratoconus and other corneal ectatic disorders. This data will be used to develop and refine a methodology for designing custom-fitted scleral contact lenses with embedded active light management technology. The study will focus on characterizing the optical imperfections (aberrations) and corneal/scleral shape variations in this population to optimize lens design for improved vision and comfort.

DETAILED DESCRIPTION:
Keratoconus, the most common corneal ectatic disease, and other related disorders are characterized by progressive thinning and steepening of the cornea, leading to distorted vision. This study will enroll individuals with these conditions to gather detailed information about their eyes using two non-invasive imaging techniques:

Wavefront aberrometry: Measures optical imperfections (aberrations) that contribute to visual distortions like glare, halos, and reduced visual acuity. This data will help understand the specific optical challenges faced by individuals with keratoconus and inform the development of lenses that correct these aberrations.

Ocular topography: Maps the three-dimensional shape of the cornea and sclera. The study will utilize advanced topography techniques to capture a wider scan of the ocular surface than is typically available. This expanded view is crucial for designing contact lenses that conform precisely to the irregular corneal shape in keratoconus (conformal fitting).

The primary objective of this study is to gather this crucial data to inform the development of a methodology for designing a conformal, custom-fitted contact lens. This lens, being developed by Azalea Vision, will incorporate active light management technology and is intended to address the complex visual challenges experienced by individuals with keratoconus and other corneal ectatic disorders. The data collected will enable Azalea Vision to optimize lens design for improved vision, comfort, and overall quality of life for these individuals.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18y
* Provide written Informed Consent
* Diagnosed with keratoconus and/or any other type of ectatic corneal disorder
* Cornea considered to be clinically stable at the discretion of the investigator (e.g. no recent cross linking performed, no current corneal sutures, no corneal sutures recently removed).
* Willing to remove current contact lenses for a minimum of 48 hours prior to performing the pentacam AXL Wave scan, if applicable.

Note: In case only 1 eye is diagnosed with keratoconus, both eyes will be scanned, as long as none of the exclusion criteria apply to that eye

Exclusion Criteria:

* Known active disease-related ocular surface problem (i.e. microbial keratitis)
* History of ocular pathologies that might lead to incomplete/incorrect eye surface scan AND wavefront aberrometry, at the discretion of the investigator
* Use of fluorescein in the eye, within 12 hours prior to the pentacam AXL Wave scan is performed
* Contact lens refitting within one month prior to the pentacam AXL Wave scan, as this can significantly impact the corneal or scleral surface.
* Currently wearing hybrid contact lenses
* Having worn contact lenses within 48 hours prior to performing the pentacam AXL Wave scan. Note: this criteria might not be applicable yet at the time of signing ICF, but needs to be confirmed prior to performing the Pentacam AXL Wave Scan

Note: In case any of the above exclusion criteria are met in 1 eye, but not in the other, it's sufficient to perform the scan on the "non" affected eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Ocular Topography | during the Eyescan procedure
  Mapping of the ocular surface
Wavefront aberrometry | during the Eyescan procedure
  Quantification of the wavefront aberrations

SECONDARY OUTCOMES:
Ocular Topography | during the Eyescan procedure
  Description of the percentage of ocular surface mapped during topography measurement
Ocular Topography | during the Eyescan procedure
  Repeatability of topography measurements between different scans will be assessed
Ocular Topography | during the Eyescan procedure
  Quality of topography measurements based on full sequence quality specification, using the parameters embedded in the Oculus Pentacam AXL Wave
Wavefront aberrometry | during the Eyescan procedure
  Quality of aberrometric measurements based on full sequence quality specification embedded in the Oculus Pentacam AXL Wave
Anterior chamber depth | during the Eyescan procedure
  as measured by the Pentacam AXL Wave.
Axial length | during the Eyescan procedure
  as measured by the Pentacam AXL Wave
Pupillometry | during the Eyescan procedure
  measurement of pupil size during aberrometry measurement
Distribution level of keratoconus severity | during the Eyescan procedure
  using the parameters embedded in the Oculus Pentacam AXL Wave

CONTACTS AND LOCATIONS:
Overall Officials: Koppen, Prof. Dr., Principal Investigator — University Hospital, Antwerp
Locations (2):
- University Hospital Antwerp (UZA), Edegem, Belgium
- Visser Contactlenzen Brunssum, Brunssum, Netherlands

IPD SHARING:
Plan to Share IPD: No
This study will be registered in a public trial register (clinicaltrials.gov) prior to inclusion of the first subject. The content - including the participating Principal Investigators and Clinical Study Sites - will be updated throughout the conduct of the study. Results information from this study will be submitted to the public trial register.